CLINICAL TRIAL: NCT05352607
Title: Effect of Transcutaneous Electrical Nerve Stimulation (TENS) on Upper Limb Spasticity in Adult Patients With Spastic Cerebral Palsy: A Randomized Control Trial
Brief Title: Effect of Transcutaneous Electrical Nerve Stimulation (TENS) on Spasticity in Adult Patients With Spastic Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reem Alharthi (Other)
Responsible Party: Sponsor-Investigator, Reem Alharthi, Physiotherapist, Umm Al-Qura University
Organization: Umm Al-Qura University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAPO-02-K-012-2022-01-912
Record Dates: First submitted 2022-04-11; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Adult; Spasticity; Transcutaneous electrical nerve stimulation; TENS; Conventional therapy
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: There will be 2 groups one is control group will receive a conventional physiotherapy treatment and the second group will receive a conventional physiotherapy treatment plus TENS therapy.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS group (Experimental): TENS group will receive the conventional physiotherapy treatment plus TENS. TENS is most commonly used directly on affected muscles in patients with CP. The device will be used from Cosmogamma company (MIXING 2 (EVO): COMBINED THERAPY). It consists of 3 parts: the stimulator part, electrode and connected wires. Strap or plaster for electrodes adhesive with gel. Electrode diameter (6×4.5 cm). The program will be (Pain therapy - TENS - Free program - Modify -Parameter's setup).
  Parameter setup (pulse frequency= 100 Hz, pulse duration= 250 μs, time=30 minutes and the intensity according to patient to feel tingling sensation only and no muscle contraction).
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Control group (Active Comparator): The Control group will receive the conventional physiotherapy treatment for upper limb spasticity only.
  Interventions: Other: Conventional physiotherapy treatment

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Put the patient in comfort position as long sitting on bed with a supported back and a pillow under the forearm, clean the skin by alcohol swab, setup the parameter, put a gel on electrodes then placed the negative electrode (black wire) over biceps belly and positive electrode (red wire) 3 cm distally from negative electrode , turn on TENS device .
  With increase the intensity gradually until patient feel a tingling sensation (no muscle contraction) and every 10 minutes ask patient about the feeling until complete 30 minutes.
  Arms: TENS group
Other: Conventional physiotherapy treatment — Application of a hot pack for 20 minutes to enhance muscle flexibility and get overall spastic muscle relaxation. Anti-spastic muscles (elbow extensors) facilitation: tapping followed by movements (three sets of 15 repetitions per session). Hand weight-bearing with bodyweight (two 5-minute per session). Passive stretching of tight muscles (elbow flexors) is used (this must be a slow and gradual stretch for 20 seconds, followed by 20 seconds of rest, five times per session). Upper-limb active exercises should be done gradually. include (finger flexion and extension exercises, elbow and shoulder (three sets of 20 reps for each session).
  Arms: Control group

SUMMARY:
Background: Cerebral palsy (CP) is a neurodevelopmental disorder caused by damage of the developing brain and marked by impairments such as increased muscle tone. Physical therapy (PT) is an important element for spasticity management include some modalities as transcutaneous electrical nerve stimulation (TENS).

Purpose: To determine the effect of TENS on inhibition of upper limb spasticity in adult patients with spastic cerebral palsy.

Methods: Twenty-four adult spastic CP patients aged from 18 to 45 years old with grade 2 to 3 spasticity according to Modified Ashworth Scale will be randomly assigned into two equal groups: TENS group and conventional therapy group. Both groups will receive conventional therapy, while TENS group in addition will receive TENS over elbow flexors with parameter setup of (pulse frequency= 100 Hz, pulse duration= 250 μs, time=30 mints) 3 sessions per week for successive 4 weeks.

Outcome measures: Modified Ashworth scale for the spasticity and digital goniometer for elbow joint range of motion, Barthel index scale for upper limb activity of daily living. Follow-up measures will be calculated three times (preintervention, post 2 weeks, and post 4 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged from 18 to 45 years old
* Diagnosed with spastic CP (upper limb is affected)
* Elbow flexor muscles spasticity grade 2 to 3 according to Modified Ashworth Scale
* Good cognition (patient able to follow the instruction)

Exclusion Criteria:

* Patient with epilepsy
* Under antispastic medication
* Severe psychological or behavioral problem
* Sensory abnormalities
* Orthopedic surgery or severe deformities in upper limb
* Injected by botulinum toxin (botox) in the past 6 months in upper limb.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-04-03 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) to assess the muscle spasticity changes | Pre intervention ( at baseline) , post 2 weeks and post 4 weeks
  The modified Ashworth scale is the most widely used clinical instrument for determining muscle tone changes. In this study will measure the elbow flexor spasticity by 3 examiners (3 minutes rest in between), then will calculate the average. MAS grades of spasticity are as follows: 0 = normal muscle tone; 1= slight increase in muscle tone, manifested by catch and release or by minimal resistance at the end; 1+ = slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout; 2= more marked increase in muscle tone, but limb easily flexed; 3= considerable increase in muscle tone, passive movement difficult; and 4 = limb rigid in flexion or extension. According to inclusion criteria, patients with grades 2 or 3 will be enrolled , then after intervention may be this grade will be deceased ( spasticity decreased ).
Digital goniometer to assess the elbow range of motion changes | Pre intervention( at baseline), post 2 weeks and post 4 weeks
  Digital goniometer is a valid tool for assessing joint range of motion. The digital goniometer has adequate concurrent criterion-related validity and comparable inter- and intra-rater reliability to the Universal goniometer. Three examiners will measure elbow joint range of motion (from full flexion to full extension), ( passively) 3 minutes rest in between.

SECONDARY OUTCOMES:
Barthel Index to assess the activity of daily living changes | Pre intervention ( at baseline) , post 2 weeks and post 4 weeks
  The Barthel is a quick and accurate, reliable assessment of mobility and activity of daily living , that works in both skillful and unskilled hands. In this study, the investigators will choose the items related to upper limb function (feeding, bathing, grooming, dressing and toilet use) with total score 40 which indicating highest independence and 0 indicating highest dependence .

CONTACTS AND LOCATIONS:
Locations (1):
- Reem Alharthi, Ta'if, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR